CLINICAL TRIAL: NCT03944174
Title: Comparative Study Between Single Trans-sacral Screw Versus Two Iliosacral Screws in Fixation of Unstable Pelvic Fractures
Brief Title: Single Trans-sacral Screw Versus Two Iliosacral Screws
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Elhady Hassan Mohammed Ali, Physician, Assiut University
Other Study IDs: Trans-sacral screw fixation
Record Dates: First submitted 2018-10-01; First posted 2019-05-09 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single Trans-sacral Screw
  Interventions: Procedure: Fixation of unstable pelvic fractures
- Two Iliosacral Screws
  Interventions: Procedure: Fixation of unstable pelvic fractures

INTERVENTIONS:
Procedure: Fixation of unstable pelvic fractures — Percutaneous fixation of both iliac bones through the sacrum using one screw

SUMMARY:
1. To compare Single Trans-sacral screw fixation vs. two Ilio-Sacral screws fixation as regard time for starting weight bearing.
2. To compare between functional outcome using the Majeed Pelvic Score.

DETAILED DESCRIPTION:
Sacroiliac screws (SISs) have been used since Vidal et al introduced them in 1973. Since that, SIS fixation has become a common technology in fixing pelvic posterior ring injuries with important progress in the past 20 years. Currently, SIS fixation represents the only minimally invasive technique to stabilize the posterior pelvic ring. For that reason, it is steadily gaining popularity, becoming one of the most commonly used techniques. The sacrum, serving as the foundation of the spine, transmits the stress between spine and pelvis through sacroiliac joints. Thus, the goal of surgical fixation is the reconstruction of the spino-pelvic-junction to allow early weight-bearing and to facilitate nursing care, particularly for multiple injured patients.

As a result of the deforming forces acting perpendicular to the implant axis, routine ilio-sacral screws fixation may not provide adequate stabilization, especially in certain unstable injuries. Longer trans-sacral screws that traverse the entire upper sacrum and exit the contralateral iliac cortex may improve holding power and also stabilize concomitant contralateral posterior pelvic injuries. These trans-sacral screws are reliably safe to insert using routine intraoperative fluoroscopy, and they provide durable fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Unstable pelvic fractures Tile type B & C.
2. Sacral Fractures.
3. Recent trauma: less than 1 week from date of trauma.
4. Neurologically free.
5. Injury Severity Score (ISS) < 18.

Exclusion Criteria:

1. Spino-pelvic dissociation.
2. Comminuted fractures
3. Bilat. Sacral fractures.
4. Sacral insufficiency.
5. Patients with associated comorbidities "eg. uncontrolled diabetes mellitus , chronic renal failure, etc.".

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any patient between 18 and 60 years old with unstable pelvic fracture admitted to the trauma unit of Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Early painless weight bearing as tolerated measured by Visual Analogue Scale of Pain (VAS). | 2 weeks
  Assessment the ability of the patient to start weight bearing without pain as soon as possible by the Visual Analogue Scale of Pain (VAS). It is a continuous scale comprised of a horizontal or vertical line, numbered from 0 to 10 and anchored by 2 verbal descriptors "no pain and worst imaginable pain" one for each symptom extreme from which the patient shall select the degree of pain varying from no pain to worst imaginable pain.
To measure the functional outcome using Majeed Pelvic Score system | 6 weeks and 6 months
  To assess the effect of the procedure on the daily activities of the patient after pelvic fractures. A system for assessment of function after major pelvic injuries is proposed. This numerical system developed from a five-year prospective study of 60 patients. Five factors were assessed and scored: pain, standing, sitting, sexual intercourse and work performance. The total score then gave a clinical grade as excellent, good, fair or poor. The scoring system allows comparison between early and late results and also between various methods of treatment.

REFERENCES:
- See also: Visual Analogue Scale of Pain — http://www.orthopaedicscore.com/scorepages/VAS_score.html
- See also: Majeed Pelvic Score — https://online.boneandjoint.org.uk/doi/abs/10.1302/0301-620X.71B2.2925751